CLINICAL TRIAL: NCT00846053
Title: FDG-PET Imaging in Young Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Thomas Ferkol, Professor of Pediatrics, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-1219
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: In this pilot study, we examined the value of FDG-PET scans as a noninvasive measure of neutrophilic inflammation in adolescents and young adults with cystic fibrosis. All subjects underwent scans.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stable lung function (Other): * Group S (n = 14) will consist of CF patients, aged 12-21 years old, who underwent FDG-PET with stable lung function during the past 4 years, defined as less than 2% decline per year. There is no therapeutic intervention and FDG-PET scan will be performed in both cohorts.
  Interventions: Diagnostic Test: FDG-PET
- Rapidly deteriorating lung function (Other): * Group R (n = 14) will contain CF patients, aged 12-21 years old, who underwent FDG-PET with rapidly deteriorating lung function during the past 4 years with greater than 4% per year decline. There is no therapeutic intervention and FDG-PET scan will be performed in both cohorts.
  Interventions: Diagnostic Test: FDG-PET

INTERVENTIONS:
Diagnostic Test: FDG-PET — All subjects underwent FDG-PET and low-dose volumetric CT imaging. After completing a transmission scan, [18F]FDG was injected intravenously at the start of dynamic scan acquisition. Regions of interest were drawn over multiple tomographic slices to determine average whole-lung and regional lung tissue [18F] FDG uptake. Patlak graphical analysis was used to determine the rate of [18F]FDG uptake from the blood input function and lung tissue activity curves, measured as the influx constant Ki (slope of the linear regression from the Patlak plot). Corrected Ki (i.e., Ki divided by the initial volume of distribution). Lung density was calculated from the attenuation image by standard methods.

SUMMARY:
The purpose of this research is to determine how a person's lungs will uptake [18F]fluorodeoxyglucose (FDG), as measured with positron emission tomography (PET) scanning in young cystic fibrosis (CF) patients.

DETAILED DESCRIPTION:
Our recent study in CF adults, supplemented by recent pre-clinical and clinical studies by our group suggests that labeled fluorodeoxyglocose-based positron emission tomography (FDG-PET) imaging may be a valuable quantitative biomarker of lung inflammation. The proposed study would validate our earlier findings, but in a younger patient population. The implications of such a test could be highly significant for both the testing of promising new anti-inflammatory agents and for patient management decisions. To capitalize on this exciting opportunity, the critical next step is to show that we can identify a cohort of young CF patients with both stable lung function and normal (or near normal) FDG-PET imaging studies. Similar patients, then, would become the subjects for a future prospective cohort study to determine if FDG-PET imaging can in fact serve as a predictor of future changes in lung function.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cystic fibrosis
* Age 12 to 21 years old, of either gender, any race or ethnicity
* Stable recent pulmonary status (defined as no new pulmonary symptoms, new antibiotic use, or hospitalization for pulmonary symptoms for at least 1 month).
* We will permit patients treated with the macrolide antibiotic, azithromycin, to participate in this study. Azithromycin has recently become a virtual standard of care in CF, based on small but reproducible improvements in pulmonary function over 4 months of treatment with this drug. The mechanism of benefit is uncertain, but an anti-inflammatory effect has been suggested. The high prevalence of use means that a study without azithromycin would likely require a wash-out period, without data about the appropriate duration for such a wash-out, or whether inflammatory markers would reverse during that time.

Exclusion Criteria:

* Failure to obtain informed consent
* Positive pregnancy test or lactation
* Currently enrolled in another study involving radioisotopes or an investigational drug
* Recent (within 30 days of screening) hospitalization for any reason
* New antibiotic use (within 30 days of screening).
* Patient incapable of lying still and supine within the PET/computed X-ray tomography (CT) scanner for 90 minutes.
* Patient incapable of completing other testing procedures (e.g., PFT, induced sputum)
* Patient with serum glucose greater than 150 mg/dl at time of PET imaging study
* Patient incapable of fasting for 4 to 6 hrs prior to PET imaging study

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ferkol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated will be published at the end of the project, consistent with normal scientific practices. Such research data will be anonymized to prevent the disclosure of personal identifiers. In return for the use of data, investigators will acknowledge our grant number in publications and presentations, and in productivity reports on publications or funding that were derived from the project, and they will not distribute materials to third-parties without notification. There will be no charge for sharing data unless the request requires effort beyond what can be subsumed under normal project budgeted effort. If the request justifies a charge, the cost is kept to a minimum and based on actual expenses.
Supporting Information: Study Protocol
Time Frame: Research data will be made available after the main findings from the final research data set have been accepted for publication. The data will be available indefinitely thereafter.
Access Criteria: Data may be shared with collaborators as approved by the Principal Investigator based on the following criteria: scientific merit, feasibility and IRB issues, appropriateness of principal investigator qualifications, and appropriateness to the project's overall goals and themes. Approval of the relevant co-investigators will be also sought and reviewed by the principal investigators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2009-December 2012, St. Louis Children's Hospital Cystic Fibrosis Clinics (St. Louis)
Groups:
- Stable Lung Function: Group S will consist of CF patients, aged 12-21 years old, with stable lung function during the past 4 years, defined as less than 2% decline per year.
- Rapidly Decline Lung Function: Group R will contain CF patients, aged 12-21 years old, with rapidly deteriorating lung function during the past 4 years with greater than 4% per year decline.
Period: Overall Study
Arm/Group | Stable Lung Function | Rapidly Decline Lung Function
Started | 13 (No milestones. Enrollment continued until end of study.) | 8
Completed | 10 (No milestones. Enrollment continued until end of study. 21 subjects enrolled.) | 8
Not Completed | 3 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stable Lung Function: Group S (n = 14) will consist of CF patients, aged 12-21 years old, with stable lung function during the past 4 years, defined as less than 2% decline per year.
- Rapidly Declining Lung Function: Group R (n = 14) will contain CF patients, aged 12-21 years old, with rapidly deteriorating lung function during the past 4 years with greater than 4% per year decline, as defined in our previous study.
- Total: Total of all reporting groups
Arm/Group | Stable Lung Function | Rapidly Declining Lung Function | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 15
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.9) | 16.6 (2.9) | 15.5 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Kinetic Influx Constant (Ki)
Description: The whole lung kinetic influx constant (Ki) is the primary outcome measure that is derived from the time-activity curves, which are generated from regions of interest placed over the whole lungs. Therefore, a single time-activity curves from each scan is used to derive the Ki.
Time Frame: At the time of FDG scan, 1 to 2 hours
Population: CF adolescents and young adults, ages 12 to 21 years, who did not have CFRD.
Measure: Mean (Standard Deviation); unit: mL/min/mL
Groups:
- Stable Lung Function: Group S (n = 10) consisted of CF patients, aged 12-21 years old, with stable lung function during the past 4 years, defined as less than 2% decline per year.
- Rapidly Declining Lung Function: Group R (n = 8) will contain CF patients, aged 12-21 years old, with rapidly deteriorating lung function during the past 4 years
Arm/Group | Stable Lung Function | Rapidly Declining Lung Function
Number analyzed (Participants) | 10 | 8
mL/min/mL | 0.009 (0.008) | 0.013 (0.008)

2. Secondary Outcome: Sputum Neutrophil Elastase (NE) Concentration
Description: Using established techniques, functional activity of neutrophil elastase in sputum sols were measured using methoxy-succinyl-ala-ala-pro-val-nitroanilide (Elastin Products, Owensville, MO), specific peptide chromogenic substrates of the neutrophil protease
Time Frame: Sample collected within 2-hours of PET scan
Population: Not every participant in the stable lung function group could produce sputum.
Measure: Mean (Standard Deviation); unit: microgram (mcg) NE /mcg protein
Groups:
- Stable Lung Function: Group S (n = 10) consists of CF patients, aged 12-21 years old, with stable lung function during the past 4 years, defined as less than 2% decline per year.
- Rapidly Declining Lung Function: Group R (n = 8) contains CF patients, aged 12-21 years old, with rapidly deteriorating lung function during the past 4 years
Arm/Group | Stable Lung Function | Rapidly Declining Lung Function
Number analyzed (Participants) | 7 | 8
microgram (mcg) NE /mcg protein | 2179 (2046) | 1656 (926)

ADVERSE EVENTS:
Time Frame: At the time of and immediately following FDG-PET scan, an average of 2-hours
Description: No difference
Groups:
- Stable Lung Function; Rapidly Declining Lung Function: No adverse events
Arm/Group | Stable Lung Function | Rapidly Declining Lung Function
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No